CLINICAL TRIAL: NCT00364169
Title: Systematic Nursing Interventions to Reduce Postoperative Constipation After Thoracic Surgery
Brief Title: Prevention of Constipation: Systematic Nursing Interventions to Reduce Postoperative Constipation After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Institute of public health, department of nursing sciences, Århus University, Denmark (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KF 01 308399
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2008-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Postoperative Constipation
Keywords: constipation; cancer; surgery; intervention; nursing; postoperative
MeSH Terms: conditions — Constipation; Neoplasms

INTERVENTIONS:
Procedure: Degree of constipation

SUMMARY:
The purpose of the study is to reduce the incidence of postoperative constipation by systematic nurse assessment, interventions and evaluation, in the first month after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for planned lung surgery
* Patients are capable
* Able to talk and understand Danish

Exclusion Criteria:

* Patients with colostomy and / or ileostomy
* Neurological or abdominal diseases
* Feed through a tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Constipation incidence the first month after surgery

SECONDARY OUTCOMES:
Defecation pattern measured after The Bristol Stool scale.
ADL (after Sallings functional scale)

CONTACTS AND LOCATIONS:
Overall Officials: Lene S. Rasmussen, RN,Stud.-MPH, Principal Investigator — Department of Cardiothoracic Surgery, The Heart Center, University hospital, Rigshospitalet, Copenhagen, Denmark; Lene S. Rasmussen, RN,Stud.-MPH, Study Director — Department of Cardiothoracic Surgery, The Heart Center, University hospital Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Department of Cardiothoracic Surgery, The Heart Center, University hospital Rigshospitalet, Copenhagen, Denmark